CLINICAL TRIAL: NCT05927688
Title: Assessment of Physician Consideration of Electronic Patient Reported Outcomes, from Patients with Gout, Rheumatoid Arthritis, Sjogren's Syndrome or Systemic Lupus Erythematosus, on the Frequency of Therapeutic Adjustments
Brief Title: Assessment of Physician Consideration of EPRO's, from Patients with Gout, Rheumatoid Arthritis, Sjogren's Syndrome or Systemic Lupus, on the Frequency of Therapeutic Adjustments
Acronym: CAPTAIN
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8546
Record Dates: First submitted 2023-06-22; First posted 2023-07-03 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Gout; Rheumatoid Arthritis; Sjogren's Syndrome; Systemic Lupus Erythematosus
MeSH Terms: conditions — Gout; Arthritis, Rheumatoid; Sjogren's Syndrome; Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients whose physician used the electronic platform to access ePRO
  Interventions: Behavioral: Therapeutic management following access by the physician to his patient's ePROs
- Patients whose physician did not used the electronic platform and did not access ePRO
  Interventions: Behavioral: Therapeutic management following access by the physician to his patient's ePROs

INTERVENTIONS:
Behavioral: Therapeutic management following access by the physician to his patient's ePROs — Therapeutic management following access by the physician to his patient's ePROs

SUMMARY:
Inflammatory rheumatic diseases affect 1% of the population. Treatment of such diseases should be based on disease activity, safety issues and other patient characteristics such as comorbidities (EULAR, 2022), leading to a higher risk of cardiovascular diseases. To this end, the general treat-to-target approach, as recommended in the EULAR guidance, may require several successive treatment lines based on updates to the patients' profile and close monitoring as the keystone of its implementation.

Regular feedback from patients could be used to fuel such strategies. This feedback can be collected using an ePRO (electronic Patient Reported Outcome). The purpose of this study is therefore to assess patient management using the information provided by patients through e-PROs, which will transfer the data provided by the patient to the physician and will notify the investigators via email when a patient has completed a form (no data interpretation or alerts).

The hypothesis is that the more physicians are provided with insights into their patients' health, the more they will function in a treat-to-target approach and the more often they will tend to adjust their patients' treatments.

ELIGIBILITY:
Inclusion Criteria:

* Men or women of at least 18 years of age
* Diagnosed with (at least) one of the following autoimmune diseases:

  * Rheumatoid arthritis (RA) according to the 2010 EULAR/ACR classification criteria,
  * Gout according to the 2015 EULAR/ACR classification criteria,
  * Systemic lupus erythematosus according to the 2019 EULAR/ACR classification criteria
  * Sjogren's Syndrome according to the 2016 EULAR/ACR classification criteria
* According to local regulations, patient has expressed his/her non-opposition (for France) or has provided written informed consent (for Switzerland and Germany) to participate in the study
* Patient has access to the internet, a functioning email address and a mobile phone number
* Patient physically and mentally able to use a computer tool connected to the Internet
* Only in Switzerland & Germany : patient is covered by a health insurance plan

Exclusion Criteria:

* Any neurodegenerative disease that alters cognitive faculties
* Refractory cancer
* Patients who do not have access to the Internet and/or do not master its use in the context of this protocol
* Unwillingness or inability to adhere to study protocol (language barriers, cognitive disorders…) Subject who is compulsorily detained for psychiatric treatment
* Patient who cannot be followed for 2 years by the investigating physician
* Patient over the age of legal majority who is protected, or deprived of liberty by judicial or administrative decision (vulnerable subject)
* Patient with an estimated life expectancy shorter than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with Gout, Rheumatoid arthritis, Sjogren's syndrome or Systemic lupus erythematosus
Sampling Method: Probability Sample
Enrollment: 352 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Frequency of therapeutic adjustments | 12 months
  To assess the relationship between the frequency of therapeutic adjustments over a 12-month period made by rheumatologists who were provided regular patient reported outcomes (PROs) and their use of an electronic platform providing them with these data.

SECONDARY OUTCOMES:
Frequency of therapeutic adjustments | 6 months
  To assess the relationship between the frequency of therapeutic adjustments over a 6-month period made by rheumatologists who were provided regular patient reported outcomes (PROs) and their use of an electronic platform providing them with these data.
Frequency of therapeutic adjustments | 24 months
  To assess the relationship between the frequency of therapeutic adjustments over a 24-month period made by rheumatologists who were provided regular patient reported outcomes (PROs) and their use of an electronic platform providing them with these data.
Frequency of flares and exacerbation | Day 1
  To assess the fluctuation of disease activity and flares - as perceived by the patient
Frequency of flares and exacerbation | 6 months
  To assess the fluctuation of disease activity and flares - as perceived by the patient
Frequency of flares and exacerbation | 12 months
  To assess the fluctuation of disease activity and flares - as perceived by the patient
Frequency of flares and exacerbation | 24 months
  To assess the fluctuation of disease activity and flares - as perceived by the patient
RAPID 3 (Routine Assessment of Patient Index Data 3) questionnaire to measure the disease score | Day 1
  To assess the overall health of patients
RAPID 3 (Routine Assessment of Patient Index Data 3) questionnaire to measure the disease score | 6 months
  To assess the overall health of patients
RAPID 3 (Routine Assessment of Patient Index Data 3) questionnaire to measure the disease score | 12 months
  To assess the overall health of patients
RAPID 3 (Routine Assessment of Patient Index Data 3) questionnaire to measure the disease score | 24 months
  To assess the overall health of patients
HAQ score (Health Assessment Questionnaire) for health assessment | Day 1
  To assess the overall health of patients
HAQ score (Health Assessment Questionnaire) for health assessment | 6 months
  To assess the overall health of patients
HAQ score (Health Assessment Questionnaire) for health assessment | 12 months
  To assess the overall health of patients
HAQ score (Health Assessment Questionnaire) for health assessment | 24 months
  To assess the overall health of patients
IPAQ score (International Physical Activity Questionnaire) to measure physical activity | Day 1
  To assess patient's physical activity over time
IPAQ score (International Physical Activity Questionnaire) to measure physical activity | 6 months
  To assess patient's physical activity over time
IPAQ score (International Physical Activity Questionnaire) to measure physical activity | 12 months
  To assess patient's physical activity over time
IPAQ score (International Physical Activity Questionnaire) to measure physical activity | 24 months
  To assess patient's physical activity over time
PEPPI score (Perceived efficacy in patient-physician interactions) | 6 months
  To assess the patient-physician relationship
PEPPI score (Perceived efficacy in patient-physician interactions) | 12 months
  To assess the patient-physician relationship
PEPPI score (Perceived efficacy in patient-physician interactions) | 18 months
  To assess the patient-physician relationship
PEPPI score (Perceived efficacy in patient-physician interactions) | 24 months
  To assess the patient-physician relationship
Number of times patients logged in to the platform | 6 months
  To assess the use of the patient portal by patients and associated satisfaction
Number of times patients logged in to the platform | 12 months
  To assess the use of the patient portal by patients and associated satisfaction
Number of times patients logged in to the platform | 24 months
  To assess the use of the patient portal by patients and associated satisfaction
Number of times physicians logged in to the platform | 6 months
  To assess the viewing of patient-reported data by physicians
Number of times physicians logged in to the platform | 12 months
  To assess the viewing of patient-reported data by physicians
Number of times physicians logged in to the platform | 24 months
  To assess the viewing of patient-reported data by physicians

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Strasbourg, Strasbourg, France